CLINICAL TRIAL: NCT04426838
Title: Cognitive Behavioral Therapy for Insomnia for the Dementia Caregiving Dyad
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Alzheimer's Association (Other)
Responsible Party: Principal Investigator, Glenna Brewster, Assistant Professor, Emory University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00115210
Record Dates: First submitted 2020-06-09; First posted 2020-06-11 (Actual); Last update posted 2023-03-20 (Actual); Status verified 2023-03

CONDITIONS: Cognitive Impairment; Dementia
Keywords: Cognitive behavioral therapy for insomnia; Insomnia; Caregiver; Cognitive impairment
MeSH Terms: conditions — Cognitive Dysfunction; Dementia; Sleep Initiation and Maintenance Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: 40 dyads of people living with dementia (PLwD) and their caregivers will be enrolled to participate in the behavioral intervention together.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PLwD Cognitive Behavioral Therapy for Insomnia (CBTi) (Experimental): Persons living with dementia in a dyad receiving the CBTi intervention in a videoconferencing format.
  Interventions: Behavioral: Cognitive Behavioral Therapy for Insomnia (CBTi) via Videoconference
- Caregiver Cognitive Behavioral Therapy for Insomnia (CBTi) (Experimental): Caregivers in a dyad receiving the CBTi intervention in a videoconferencing format.
  Interventions: Behavioral: Cognitive Behavioral Therapy for Insomnia (CBTi) via Videoconference

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy for Insomnia (CBTi) via Videoconference — The CBTi protocol will include stimulus control, sleep compression, relaxation, sleep hygiene, and cognitive restructuring which will be done over 4 weeks with one session weekly delivered via videoconference.

SUMMARY:
Disturbed sleep is stressful to persons living with dementia (PLwD) and their caregivers. It contributes to earlier placement of the PLwD in nursing homes and increase the risk for many psychological and cognitive health issues and poor quality of life for both the PLwD and the caregivers. Given the potential harmful side effects of medications, non-medication alternatives, such as Cognitive Behavioral Therapy for Insomnia (CBTi), may be safer to improve disturbed sleep in this population. CBTi which includes stimulus control, sleep compression, relaxation, sleep hygiene, and cognitive restructuring, is effective and has durable and sustained effects on sleep outcomes over the long-term. CBTi has improved sleep disturbances in PLwD and their caregivers, separately. Since disturbed sleep in the PLwD-caregiver dyad is bidirectional and interdependent, targeting the pair as a unit for intervention has the potential to lead to improved sleep and health outcomes for both persons. There is no current published research on CBTi when the PLwD and their caregivers receive the intervention at the same time; as a result, the researchers will examine the 1) feasibility; 2) acceptability; and 3) preliminary efficacy of 4-week CBTi intervention for community-dwelling PLwD and their caregivers who are both experiencing sleep disturbances. Forty PLwD-caregiver dyads will receive CBTi via videoconferencing sessions. Preliminary efficacy of the intervention will be assessed using objective (actigraphy) and subjective sleep quality measures. In addition, semi-structured interviews will be conducted to examine the acceptability and satisfaction with the intervention.

DETAILED DESCRIPTION:
Up to 71% of the persons living with dementia (PLwD) and 70% of their caregivers experience sleep disturbances, which are distressing for both the PLwD and their caregivers. Specifically, PLwD often experience restlessness and fragmented sleep, which in turn can affect caregivers' sleep patterns leading to multiple nightly awakenings, shorter sleep duration, and/or inconsistent sleep-wake times. These disturbances increase the risk for a myriad of psychological, cognitive, behavioral, and physiological health issues and poor quality of life for the dyad. Given the interdependence of the dyadic sleep disturbances and the negative health consequences of sleep disturbances on the dyad, there is a critical need to develop and provide effective interventions to improve their sleep. Pharmacologic treatment often results in potential harmful side effects like falls and cognitive decline; therefore, non-pharmacologic approaches are recommended for this population.

Cognitive behavioral therapy for insomnia (CBTi), a non-pharmacologic intervention that has demonstrated effectiveness for improving sleep disturbances in multiple populations, is delivered in various formats including face-to-face and videoconferencing. Individually, PLwD and caregivers have successfully deployed behavioral sleep techniques, resulting in improved sleep quality. However, there is no current published research on CBTi completed simultaneously by the PLwD-caregiver dyad, and that is exactly what the researchers of this study seek to do with early-stage individuals and their caregivers. The researchers premise this effort on the notion that a dyadic intervention can use early-stage individuals' retained capacity for communication and comprehension to establish in-the-moment agreements about strategies the caregiver can employ to enact and facilitate positive sleep behaviors in the PLwD and to pair that with acquired strategies to engender his/her own positive sleep behaviors.

This project seeks to gather formative and preliminary data on CBTi delivered simultaneously to the PLwD-caregiver dyad. The researchers will use a quantitative, descriptive approach to determine the feasibility, acceptability, and preliminary efficacy of a 4-session CBTi intervention administered to 40 PLwD-caregiver dyads via videoconferencing sessions who will receive the intervention as a unit. Objective and subjective sleep, depressive symptoms, and cognitive health data will be collected at baseline, and 1 week and 3 months post-completion of the intervention.

In community-dwelling PLwD and their caregivers where both persons in the dyad self-report sleep disturbances, the specific aims for this study are:

1. Assess the feasibility of a video conferencing dyad-based CBTi intervention.
2. Evaluate the acceptability of a video conferencing dyad-based CBTi intervention.
3. Examine the preliminary efficacy of video conferencing CBTi intervention on sleep quality outcomes including sleep efficiency and perceived sleep quality.

ELIGIBILITY:
Inclusion Criteria for the PLwD

* Caregiver-reported diagnosis of cognitive impairment and Alzheimer's disease and related dementias (ADRD)
* Co-residence with the caregiver in the community
* Montreal Cognitive Assessment (MOCA) score between 12 and 25
* Stable dose of psychotropic medications, anti-dementia, sedatives/hypnotics, or opioids in the past 90 days
* Presence of sleep problems determined by using the proxy-rated Sleep Disorders Inventory (presence of at least one sleep disturbance symptom of moderate severity)

Inclusion Criteria for the Caregiver

* Informal caregivers (family/friends) of co-residing PLwD
* Providing unpaid assistance, on average 20 hours weekly, for a person in the early stage of illness who is community-dwelling
* Presence of sleep problems: sleep onset latency or wake after sleep onset more than 30 minutes more than 3 nights weekly

Inclusion Criteria for the Dyad

* Tolerate and agrees to wear wrist actigraph
* Be able to read, speak and understand English
* Have no uncorrectable vision or hearing deficits that might impede participation

Exclusion Criteria for the PLwD

* None

Exclusion Criteria for the Caregivers

* Moderate to severe cognitive impairment defined as MoCA score <17
* Current sedative-hypnotic or other sleep aid use on a regular or as needed schedule within the prior three months
* Presence of an acute medical or psychiatric condition which would interfere with the subject's ability to realistically follow the study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2020-09-30 (Actual); Primary Completion 2023-03-10 (Actual); Study Completion 2023-03-10 (Actual)

PRIMARY OUTCOMES:
Change in Adherence with Study Interventions | Weeks 1, 2, 3, 4
  Feasibility of the interventions will be assessed with rates of adherence to the study components weekly and over the 4 weeks
Percent Attrition from the Study | Week 4
  Feasibility of the interventions will be assessed with the percent of participants leaving the study over the 4 week intervention.
Acceptability the Intervention | Week 5 (1 week post-intervention)
  Acceptability of the interventions will be assessed with a qualitative interview with caregivers after completing the intervention. There is not a summary score for the open-ended questions asked during the interview.

SECONDARY OUTCOMES:
Change in Sleep Disorders Inventory (SDI) - Frequency Score | Baseline, Week 5 (1 week post-intervention), Month 4 (1 month post-intervention)
  The SDI asks caretakers to report the frequency that eight symptoms of insomnia have been exhibited by the PLwD in the past two weeks. Responses range from 0 to 4 where 0 = not present and 4 = every night. Total frequency scores range from 0 to 32 with higher scores indicating more frequent symptoms of insomnia.
Change in Sleep Disorders Inventory (SDI) - Severity Score | Baseline, Week 5 (1 week post-intervention), Month 4 (1 month post-intervention)
  The SDI asks caretakers to report the severity of eight symptoms of insomnia being exhibited by the PLwD in the past two weeks. Responses range from 0 to 3 where 0 = not present and 3 = marked. Total frequency scores range from 0 to 24 with higher scores indicating more severe symptoms of insomnia.
Change in Sleep Disorders Inventory (SDI) - Caregiver Distress Score | Baseline, Week 5 (1 week post-intervention), Month 4 (1 month post-intervention)
  The SDI asks caretakers to report the amount of distress they are experiencing due to eight symptoms of insomnia being exhibited by the PLwD in the past two weeks. Responses range from 0 to 5 where 0 = not at all and 5 = extremely. Total frequency scores range from 0 to 40 with higher scores indicating more severe caregiver distress.
Change in Insomnia Severity Index Score | Baseline, Week 5 (1 week post-intervention), Month 4 (1 month post-intervention)
  The Insomnia Severity Index includes 7 questions asking about insomnia during the past two weeks. Responses are given on a scale from 0 to 4 where 0 = no problems and 4 = the most extreme problems. Total scores range from 0 to 28 where higher scores indicate greater problems with insomnia.
Change in 12-Item Short Form-12 (SF-12v2) Health Survey Score | Baseline, Week 5 (1 week post-intervention), Month 4 (1 month post-intervention)
  The SF-12 Health Survey includes 12 items asking respondents how they have been feeling and activities they are doing. Physical and mental health composite scores are computed and range from 0 to 100 where 100 is the highest level of health. The computed composite scores can be compared with a national norm with a mean of 50 and a standard deviation of 10.
Change in Center for Epidemiologic Studies Depression Scale (CES-D) Score | Baseline, Week 5 (1 week post-intervention), Month 4 (1 month post-intervention)
  The CES-D includes 20 items asking respondents how frequently they felt symptoms of depression during the past week. Responses are given on a scale from 0 to 3 where 0 = rarely or none of the time and 3 = most or all of the time. Certain items are reverse scored so that lower scores equate to lower symptom frequency. Total scores range from 0 to 60 with higher scores indicating greater symptoms of depression.
Change in Sleep Duration | Baseline (for two weeks prior to the intervention), Day 1 through Week 4
  Participants will wear an actigraph for two weeks before the intervention starts and for the duration of the intervention. Sleep duration (minutes per night) will be assessed with actigraphy.
Change in Sleep Fragmentation Index | Baseline (for two weeks prior to the intervention), Day 1 through Week 4
  Participants will wear an actigraph for two weeks before the intervention starts and for the duration of the intervention. The sleep fragmentation index (number of awakenings and sleep stage shifts divided by sleep time) will be assessed with actigraphy.
Change in Sleep Onset Latency | Baseline (for two weeks prior to the intervention), Day 1 through Week 4
  Participants will wear an actigraph for two weeks before the intervention starts and for the duration of the intervention. Sleep onset latency (the length of time, in minutes, that it takes to transition from wakefulness to sleep) will be assessed with actigraphy.
Change in Wake After Sleep Onset | Baseline (for two weeks prior to the intervention), Day 1 through Week 4
  Participants will wear an actigraph for two weeks before the intervention starts and for the duration of the intervention. Wake after sleep onset (periods of wakefulness occurring after sleep onset) will be assessed with actigraphy.
Change in Bed Time | Baseline (for two weeks prior to the intervention), Day 1 through Week 4
  Participants will wear an actigraph for two weeks before the intervention starts and for the duration of the intervention. Bed time will be assessed with actigraphy.
Change in Wake Time | Baseline (for two weeks prior to the intervention), Day 1 through Week 4
  Participants will wear an actigraph for two weeks before the intervention starts and for the duration of the intervention. Wake time will be assessed with actigraphy.

CONTACTS AND LOCATIONS:
Overall Officials: Glenna Brewster, PhD, RN, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Emory University, Atlanta, Georgia
  - Goizueta Alzheimer's Disease Research Center, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: No